CLINICAL TRIAL: NCT04620577
Title: The Influence of Antibiotics on the Incidence of Biliary Tract Infections After PTCD for Malignant Obstructive Jaundice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xian-Jun Yu (Other)
Responsible Party: Sponsor-Investigator, Xian-Jun Yu, President of Shanghai Pancreatic Cancer Institute, Fudan University
Organization: Fudan University (Other)
Other Study IDs: FudanU
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: The Influence of Antibiotics on the Incidence of Biliary Tract Infections After PTCD for Malignant Obstructive Jaundice
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antibiotic group: Infusion of ceftriaxone sodium needle (2g, solvent 100ml normal saline) within 1h before and 12h after PTCD.
  Interventions: Other: antibiotic
- No-antibiotic group: Infusion of Normal saline within 1h before and 12h after PTCD.
  Interventions: Other: antibiotic

INTERVENTIONS:
Other: antibiotic — normal saline

SUMMARY:
To investigate the influence of antibiotics on the incidence of biliary tract infections after PTCD for malignant obstructive jaundice.

DETAILED DESCRIPTION:
This project designed a large-scale, single-center, prospective randomized controlled clinical trial to explore the impact of antibiotics on the incidence of biliary tract infections after PTCD with malignant obstructive jaundice. This study will provide evidence-based medical evidence for the need for routine use of antibiotics to prevent biliary tract infections after PTCD with malignant obstructive jaundice, and provide references for clinicians to prevent patients from PTCD infections.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old;
2. ECOG score 0-1 before operation;
3. Patients diagnosed as pancreatic head cancer and periampullary cancer according to preoperative imaging, including ampullary cancer, extrahepatic bile duct cancer and duodenal papillary cancer;
4. Bilirubin>200 mmol/L before PTCD , and the duration of PTCD continuous drainage >2 weeks;
5. Volunteer to participate and sign the informed consent form;

Exclusion Criteria:

1. Decompensated liver cirrhosis, acute and chronic hepatitis and other diseases before surgery;
2. A history of other malignant tumors before surgery;
3. Duration of preoperative PTCD drainage<2 weeks;
4. Jaundice caused by other reasons besides cancer around the ampulla and cancer of the head of the pancreas;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with periampullary carcinoma and pancreatic head carcinoma who received PTCD drainage.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of patients with biliary tract infection after surgery | October 2020 to June 2023
  Incidence of patients with biliary tract infection after surgery

SECONDARY OUTCOMES:
Decline rate of bilirubin in patients after PTCD | October 2020 to June 2023
  Decline rate of bilirubin in patients after PTCD

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided